CLINICAL TRIAL: NCT05187611
Title: Conduction System Pacing vs Biventricular Resynchronization Therapy in Systolic Dysfunction and Wide QRS: CONSYST-CRT Randomized Clinical Trial.
Brief Title: Conduction System Pacing vs Biventricular Resynchronization Therapy in Systolic Dysfunction and Wide QRS: CONSYST-CRT.
Acronym: CONSYST-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONSYST-CRT.
Record Dates: First submitted 2021-12-19; First posted 2022-01-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Resynchronization Therapy; Conduction System Pacing
Keywords: Resynchronization Therapy; Biventricular pacing; Conduction system pacing
MeSH Terms: interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: The first 70 patients have been recruited in the context of the LEVELAT study (ClinicalTrials.gov Identifier: NCT04054895)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conduction system pacing (Experimental): Pacing the His-Purkinje system.
  Crossover to biventricular pacing was allowed in case of failed conduction system pacing: failed His bundle pacing and failed Left bundle branch pacing (high thresholds (>3.5V / 1ms); no left bundle branch pacing criteria; no left bundle branch correction).
  Electrocardiographic optimization allowed in order to obtain the narrowest QRS.
  Interventions: Device: Conduction system pacing
- Biventricular pacing (Active Comparator): Pacing from the right ventricular and coronary sinus leads. Electrocardiographic optimization with fusion-optimized intervals.
  Crossover from biventricular pacing to conduction system pacing will be allowed in the following situations: coronary sinus cannot be cannulated; no lateral or posterolateral branches; or phrenic stimulation.
  Interventions: Device: Biventricular pacing

INTERVENTIONS:
Device: Conduction system pacing — Lead placed in the His-Purkinje system in order to achieve QRS shortening.
  Arms: Conduction system pacing
Device: Biventricular pacing — Lead is placed in a tributary of the coronary sinus.
  Arms: Biventricular pacing

SUMMARY:
Conduction system pacing vs biventricular resynchronization therapy in systolic dysfunction and wide QRS (CONSYST-CRT randomized clinical trial) is a non-inferiority trial that aims to study the composite endpoint consisting of all-cause mortality, cardiac transplant, heart failure hospitalizations, and left ventricular ejection fraction (LVEF) improvement <5 points.

DETAILED DESCRIPTION:
To date, studies have shown that conduction system pacing could get similar clinical and echocardiographic responses to those obtained with biventricular therapy.

This study will randomize 130 patients to a strategy of biventricular pacing versus conduction system pacing.

CONSYST-CRT study will analyze the following parameters in the 2 groups: left ventricular ejection fraction, ventricular volumes, echocardiographic response (>=15% decrease in left ventricular end-systolic volume), NYHA functional class, heart failure hospitalization, all-cause mortality, cardiac transplant, QRS shortening, echocardiographic asynchrony (septal flash).

Clinical, electrocardiographic, echocardiographic follow-up will be performed for 1 year.

The first 70 patients have been recruited in the context of the LEVELAT study (ClinicalTrials.gov Identifier: NCT04054895)

ELIGIBILITY:
Inclusion Criteria:

* The patient must indicate their acceptance to participate in the study by signing an informed consent document.
* The patient must be ≥ 18 years of age.
* Left bundle branch block, QRS ≥130 and LVEF <=35%. No indication of stimulation for AV block.
* Non-left bundle branch block, QRS ≥150 and LVEF <=35%.
* Patients with indication of resynchronization therapy for ventricular dysfunction (LVEF <40%) and indication of cardiac pacing for AV block.
* LVEF <=35% in NYHA class III or IV if they are in atrial fibrillation and have intrinsic QRS >=130 ms, provided a strategy to ensure biventricular capture is in place.

Exclusion Criteria:

* Myocardial infarction, unstable angina or cardiac revascularization during the previous 3 months.
* Pregnancy.
* Participating currently in a clinical investigation that includes an active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Composite end-point: all-cause mortality, cardiac transplant, heart failure hospitalization, and left ventricular ejection fraction (LVEF) improvement <5 points. | 12 months
  Non inferiority margin 10%.

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction. | 6 months; 12 months
  Non inferiority margin 2.5%
Change in left ventricular end-systolic volume. | 6 months; 12 months
  Non inferiority margin 3%
Echocardiographic response (>=15% decrease in left ventricular end-systolic volume). | 6 months; 12 months
  Non inferiority margin 10%
Hospitalization due to heart failure, mortality or cardiac transplant (combined endpoint) | 6 months; 12 months
  Non inferiority margin 10%
QRS shortening | Post-implantation (Electrophysiology Lab)
  Non inferiority margin 12ms
Correction of septal flash | 15 days; 6 months; 12 months
  Non inferiority margin 0.5mm
Change in NYHA functional class | 6 months; 12 months
  NYHA functional class I, II, III, IV.

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Mont, MD, PhD, Study Director — Hospital Clinic of Barcelona; Jose M Tolosana, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Margarida Pujol Lopez, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Lluís Mont, Barcelona, Spain

REFERENCES:
- [Derived] Pujol-Lopez M, Graterol FR, Borras R, Garcia-Ribas C, Guichard JB, Regany-Closa M, Jimenez-Arjona R, Niebla M, Poza M, Carro E, Castel MA, Arbelo E, Porta-Sanchez A, Sitges M, Roca-Luque I, Doltra A, Guasch E, Tolosana JM, Mont L. Clinical Response to Resynchronization Therapy: Conduction System Pacing vs Biventricular Pacing: The CONSYST-CRT Trial. JACC Clin Electrophysiol. 2025 Aug;11(8):1820-1831. doi: 10.1016/j.jacep.2025.03.024. Epub 2025 May 14. PMID 40372330